CLINICAL TRIAL: NCT01440699
Title: Phase I Study of Dose Escalation of Human Allogenic Adipose-derived Stem Cells (ALLO-ASC) to Evaluate Safety and Efficacy in Patients With Crohn's Fistula
Brief Title: Study of Allogenic Adipose-derived Stem Cells in Crohn's Fistula
Acronym: ALLO-ASC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-101
Record Dates: First submitted 2011-09-19; First posted 2011-09-26 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2011-09

CONDITIONS: Crohn
Keywords: Crohn's fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): For ALLO-ASC 1xE7 cells/ml,3 patients are to be enrolled. If there is no safety issue, 3 more patients will be enrolled to be treated with ALLO-ASC 3xE7 cells/ml.
  Interventions: Biological: Allogenic human adipose-derived stem cells

INTERVENTIONS:
Biological: Allogenic human adipose-derived stem cells — ALLO-ASC 1xE7 cells/mL is injected once along the fistula. If there is no safety issue for 4 weeks, 3 more people could be enrolled who are subject to ALLO-ASC 3xE7 cells/mL.
  Other Names: ALLO-ASC

SUMMARY:
Adipose-derived stem cells have properties of differentiation to various types of cells, immunomodulatory effects. adipose-derived stem cells (ASCs) show also low immunogenicity.

Anterogen has developed ANTG-ASC(Autologous ASC) which has shown good efficacy and safety in Phase I and II study on the patients with Crohn's fistula.

However, Crohn's patients are sometimes not fat enough to extract fat tissue for culturing ASCs. Therefore the investigators have planned to study allogenic ASCs for safety and efficacy in patients with Crohn's fistula.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Crohn's disease
* Crohn's fistula which has been lasted at least for 3 months
* Negative for beta-HCG pregnancy test

Exclusion Criteria:

* Medical history with Variant Creutzfeldt Jacobs Disease
* Allergic to anesthetics or bovine protein or fibrin glue
* autoimmune disease other than Crohn's disease
* Infectious disease
* Sepsis or active tuberculosis
* pregnant or breast feeding woman
* Inflammatory Bowel disease other than Crohn's disease
* active crohn's disease with CDAI score > 200
* malignant tumor
* fistula's diameter > 2 cm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10-11 (Actual); Study Completion 2012-11-08 (Actual)

PRIMARY OUTCOMES:
General safety (Laboratory screening, adverse effects, immunological response, local tolerance) | Week8

SECONDARY OUTCOMES:
Proportion of patients with sustained efficacy | Month 8
  Proportion of patients with more than 50% healed fistula at Month 8 Following up whether there is a recurrence at Month 8
Proportion of patients with adverse effects | at month 8
  Evaluate the safety at 8 months whether any kind of AE occurs.

CONTACTS AND LOCATIONS:
Overall Officials: TI Kim, MD, PhD, Principal Investigator — Yeonsei Medical Center
Locations (3):
- South Korea (3):
  - Keonghee Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yeonsei Medical Center, Seoul